CLINICAL TRIAL: NCT01994460
Title: Substitution of Ethambutol With Linezolid During the Intensive Phase of Treatment of Pulmonary Tuberculosis: A Prospective, Multicenter, Randomized, Open-label Phase II Trial
Brief Title: Linezolid Instead of Ethambutol in Treatment of Drug-susceptible Tuberculosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); SMG-SNU Boramae Medical Center (Other); Seoul National University Bundang Hospital (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J-1310-026-523
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Pulmonary Tuberculosis Without Resistance to Rifampicin
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Linezolid; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (control arm) (Active Comparator): Standard treatment for drug-sensitive pulmonary TB using isoniazid (6 months), rifampicin (6 months), pyrazinamide (2 months), and ethambutol (2 months)
  Interventions: Drug: Ethambutol
- Arm 2 (experimental arm 1) (Experimental): Isoniazid (6 months), rifampicin (6 months), pyrazinamide (2 months), and linezolid (600 mg/day, 2 weeks)
  Interventions: Drug: Linezolid
- Arm 3 (experimental arm 2) (Experimental): Isoniazid (6 months), rifampicin (6 months), pyrazinamide (2 months), and linezolid (600 mg/day, 4 weeks)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid
  Arms: Arm 2 (experimental arm 1); Arm 3 (experimental arm 2)
Drug: Ethambutol
  Arms: Arm 1 (control arm)

SUMMARY:
The current standard short-course treatment for pulmonary TB requires 6 months to complete. This long duration of treatment increases the likelihood of side effects while decreasing patients' adherence to anti-TB drugs. Linezolid showed considerable efficacy against refractory multidrug-resistant TB. Considering the marked anti-TB effects of linezolid as well as the possible adverse effects of its long-term use, it is rational to use linezolid instead of ethambutol for the first 4 weeks of treatment for drug-susceptible pulmonary TB. Through randomized controlled trial, the investigators will evaluate the hypothesis that the use of linezolid instead of ethambutol will increase the sputum culture conversion rate by 15% after 2 months of treatment. Patients with TB without resistance to rifampicin will be randomized to the following three arms at a 1:1:1 ratio: Arma 1 (control arm), Arm 2 (linezolid for 2 weeks instead of ethambutol), Arm 3 (linezolid for 4 weeks instead of ethambutol)Primary outcome will be sputum culture conversion rate after 2 months of treatment (liquid media).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged from 20 to 80 years (20- and 80-year-old patients can participate).
* Documented sputum Xpert MTB/RIF assay-positive pulmonary TB at screening.
* On current TB therapy (if any) for ≤14 days at the time of enrollment.

Exclusion Criteria:

* Patients with HIV/AIDS.
* Females of childbearing potential, who are pregnant, breastfeeding, or unwilling to avoid pregnancy.
* Any of the following:

  i.Absolute neutrophil count of <2000 cells/mL. ii.White blood cell count (WBC) of <3000/μL. iii.Hemoglobin concentration of <7.0 g/dL. iv.Serum creatinine level of >2.0 mg/dL. v.Aspartate aminotransferase (AST or SGOT) of >100 IU/L. vi.Alanine aminotransferase (ALT or SGPT) of >100 IU/L. vii.Total bilirubin level of >2.0 mg/dL. viii.History of optic neuritis or peripheral neuropathy. ix.Other significant laboratory abnormalities (i.e., absolute neutrophil count, creatinine level).

  x.The need for ongoing therapy with SSRIs, tricyclic antidepressants, serotonin 5-HT1 receptor agonists (triptans), meperidine, buspirone, monoamine oxidase inhibitors (MAOIs), sympathomimetic agents (e.g., pseudoephedrine), vasopressive agents (e.g., epinephrine, norepinephrine), or dopaminergic agents (e.g., dopamine, dobutamine).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Sputum culture conversion rate on liquid media | after 2 months of treatment

SECONDARY OUTCOMES:
Sputum culture conversion rate on solid media | after 2 months of treatment
Time to sputum culture conversion (liquid and solid media) | During 6 months of treatment
Cure rate | After 6 months of treatment
Treatment success rate | after 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam, Kyunggi
  - National Medical Center, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul

REFERENCES:
- [Derived] Lee JK, Lee JY, Kim DK, Yoon HI, Jeong I, Heo EY, Park YS, Jo YS, Lee JH, Park SS, Park JS, Kim J, Lee SM, Joh JS, Lee CH, Lee J, Choi SM, Park JH, Lee SH, Cho YJ, Lee YJ, Kim SJ, Kwak N, Hwang YR, Kim H, Ki J, Lim JN, Choi HS, Lee M, Song T, Kim HS, Han J, Ahn H, Hahn S, Yim JJ. Substitution of ethambutol with linezolid during the intensive phase of treatment of pulmonary tuberculosis: a prospective, multicentre, randomised, open-label, phase 2 trial. Lancet Infect Dis. 2019 Jan;19(1):46-55. doi: 10.1016/S1473-3099(18)30480-8. Epub 2018 Nov 23. PMID 30477961
- [Derived] Lee JY, Kim DK, Lee JK, Yoon HI, Jeong I, Heo E, Park YS, Lee JH, Park SS, Lee SM, Lee CH, Lee J, Choi SM, Park JS, Joh JS, Cho YJ, Lee YJ, Kim SJ, Hwang YR, Kim H, Ki J, Choi H, Han J, Ahn H, Hahn S, Yim JJ. Substitution of ethambutol with linezolid during the intensive phase of treatment of pulmonary tuberculosis: study protocol for a prospective, multicenter, randomized, open-label, phase II trial. Trials. 2017 Feb 13;18(1):68. doi: 10.1186/s13063-017-1811-0. PMID 28193240